CLINICAL TRIAL: NCT06121843
Title: A Phase 1, Multicenter, Open-label Study to Evaluate the Safety and Preliminary Efficacy of Arlocabtagene Autoleucel (BMS-986393) in Novel Combinations in Participants With Relapsed and/or Refractory Multiple Myeloma and Determine the Recommended Dose for Each Add-on Investigational Component
Brief Title: A Study to Evaluate the Safety, Effectiveness and Tolerable Dose of Arlocabtagene Autoleucel (BMS-986393) in Novel Combinations in Participants With Relapsed and/or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA088-1005
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: BMS-986393; Relapsed Multiple Myeloma; Refractory Multiple Myeloma; First-in-human; Alnuctamab; Mezigdomide; Iberdomide; CC-95266; GPRC5D; GPRC5D CAR T; Cell Therapy; CAR T cell therapy; Combination therapy; elranatamab; arlocabtagene autoleucel; arlo-cel
MeSH Terms: conditions — Multiple Myeloma | interventions — iberdomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: BMS-986393 + Alnuctamab (Experimental)
  Interventions: Drug: BMS-986393; Drug: Alnuctamab
- Arm B: BMS-986393 + Mezigdomide (Experimental)
  Interventions: Drug: BMS-986393; Drug: Mezigdomide
- Arm C: BMS-986393 + Iberdomide (Experimental)
  Interventions: Drug: BMS-986393; Drug: Iberdomide
- Arm D: BMS-986393 + Elranatamab (Experimental)
  Interventions: Drug: BMS-986393; Drug: Elranatamab

INTERVENTIONS:
Drug: BMS-986393 — Specified dose on specified days
  Other Names: CC-95266; Arlocabtagene autoleucel; arlo-cel
Drug: Alnuctamab — Specified dose on specified days
  Other Names: BMS-986349; CC-93269; EM901
  Arms: Arm A: BMS-986393 + Alnuctamab
Drug: Mezigdomide — Specified dose on specified days
  Other Names: BMS-986348; CC-92480
  Arms: Arm B: BMS-986393 + Mezigdomide
Drug: Iberdomide — Specified dose on specified days
  Other Names: BMS-986382; CC-220
  Arms: Arm C: BMS-986393 + Iberdomide
Drug: Elranatamab — Specified dose on specified days
  Other Names: Elrexfio
  Arms: Arm D: BMS-986393 + Elranatamab

SUMMARY:
The purpose of this study is to establish a safe and tolerable dose of arlocabtagene autoleucel (BMS-986393) in combinations with alnuctamab, mezigdomide, iberdomide, and elranatamab in participants with relapsed and/or refractory multiple myeloma (RRMM).

ELIGIBILITY:
Inclusion Criteria:

* History of relapsed and/or refractory multiple myeloma (RRMM) treated with at least 3 (Part 1 and Part 2) or at least 1 but not greater than 3 prior anti-myeloma treatment regimens (Part 2).
* Measurable multiple myeloma (MM).
* Eastern Cooperative Oncology Group performance status of 0-1.

Exclusion Criteria:

* Prior treatment with alnuctamab (Arm A), mezigdomide (Arm B), iberdomide (Arm C), elranatamab (Arm D) or BCMA-targeting therapy (Part 2 Arms A and D).
* Prior treatment with GPRC5D-targeting therapies.

Note: Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 2 years
Incidence of serious adverse events (SAEs) | Up to 2 years
Incidence of adverse events of special interest (AESI) | Up to 2 years
Incidence of AEs leading to discontinuation | Up to 2 years
Number of Deaths | Up to 2 years
Establish recommended Phase 2 dose (RP2D) | Up to 2 years

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
Complete response rate (CRR) | Up to 2 years
Very good partial response rate (VGPRR) | Up to 2 years
Maximum observed concentration (Cmax) of arlocabtagene autoleucel | Up to 2 years
Time of maximum observed concentration (tmax) of arlocabtagene autoleucel | Up to 2 years
Area under the concentration-time curve from time 0 to 28 days [AUC (0-28D)] of arlocabtagene autoleucel | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (19):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic in Arizona - Phoenix, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northside Hospital, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Local Institution - 0009, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Local Institution - 0023, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06121843.html